CLINICAL TRIAL: NCT03914066
Title: A Group-based Treatment of Overweight and Obesity in Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We could not continue the study and include participants because of the corona pandemic.
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 267621
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-05

CONDITIONS: Overweight and Obesity
Keywords: overweight; obesity; group treatment; primary care
MeSH Terms: conditions — Overweight; Obesity | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group treatment in primary care (Experimental): The intervention is a group treatment of overweight and obesity in primary care inspired by cognitive behavioural therapy. The main goal of the group treatment is for the participants to obtain and maintain healthy lifestyle habits, with emphasis on diet and physical activity. Every group has 8-12 participants and is led by two persons; the main group leader is either a primary care nurse or a physiotherapist with special training. The groups meet six times (2 hours every time) once a month over a 6-8 month period. Every group session has a set agenda with different topics, for example a healthy diet, recommended physical activity or how to deal with setbacks. Between group sessions there are home assignments. The home assignments are followed-up at the next session and participants are encouraged to share experiences with each other in order to inspire, challenge and help fellow group participants. Data is collected prior to the start of group treatment, after 6-8 and 12 months.
  Interventions: Behavioral: A group-based treatment of overweight and obesity

INTERVENTIONS:
Behavioral: A group-based treatment of overweight and obesity — The intervention is a group treatment of overweight and obesity in primary care inspired by cognitive behavioural therapy. The main goal of the group treatment is for the participants to obtain and maintain healthy lifestyle habits, with emphasis on diet and physical activity. Every group has 8-12 participants and is led by two persons; the main group leader is either a primary care nurse or a physiotherapist with special training. The groups meet six times (2 hours every time) once a month over a 6-8 month period. Every group session has a set agenda with different topics, for example a healthy diet, recommended physical activity or how to deal with setbacks. Between group sessions there are home assignments. The home assignments are followed-up at the next session and participants are encouraged to share experiences with each other in order to inspire, challenge and help fellow group participants. Data is collected prior to the start of group treatment, after 6-8 and 12 months.

SUMMARY:
Overweight and obesity is a growing problem in the world. Today more than 50 % of all people over 18 years in Sweden are overweight or obese. Main reasons for this are changes in lifestyle habits regarding diet and physical exercise. Overweight and obesity increases risk of different diseases such as type 2 diabetes, arthrosis and cancer; it also affects quality of life. Losing 5-10 % of your body weight improves metabolic health and quality of life. Lifestyle changes are very important in order to lose weight but it can be challenging to carry through with these changes on your own without support. In the primary care in Region Orebro län a group treatment, "Step by step", has been in use since 2010. It comprises of six group sessions over 6-8 months with different themes such as diet, physical exercise and stress. Between the group sessions there are home assignments, such as writing a diet or exercise diary. This observational study will evaluate "Step by step" and the effect the group treatment has on the participants' weight, dietary habits, physical activity, quality of life, eating habits and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* BMI 30 or over
* BMI over 28 and under 30 with one or more of following: hypertension, prediabetes, type 2 diabetes, coronary heart disease, hyperlipidaemia, liver steatosis, sleep apnoea or polycystic ovary syndrome.

Exclusion Criteria:

* Severe mental illness
* Previous or present eating disorder
* Pregnancy
* Breast feeding
* Serious cancer under treatment
* Use of weight-loss drugs
* Misuse of alcohol or drugs
* Type 1 diabetes
* Not being able to speak/read/write Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Weight reduction in kg and % from baseline to 6-8 months and 12 months. | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured in kilograms

SECONDARY OUTCOMES:
Change in Dietary habits | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by a questionnaire from The National Board of Health and Welfare with 4 questions regarding how often the person eats vegetables, fruit, fish and sweets.
Change in Physical activity | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by accelerometer.
Change in general Health-related Quality of Life | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by Rand 36-item Health survey. Comprises 36 items that assess 8 health concepts: physical functioning, role limitations, social functioning, emotional wellbeing, energy/fatigue, pain and general health perceptions. Subscale scores range from 0 to 100, where higher scores represent better health status.
Change in Obesity-specific Health-related Quality of Life | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by the Obesity-Related Problems scale (OP V1.2). Comprises 8 items with a response choice from 1-4: 1 = Definitely bothered, 2 = Mostly bothered, 3 = Not so bothered and 4 = Definitely not bothered. The scores are transformed to a raw scale score that is then transformed to a 0-100 scale. A higher score indicates more psychosocial problems.
Change in Eating patterns | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by the Three-Factor Eating Questionnaire (TFEQ-R18v2). Comprises 18 items that measure 3 domains of eating behaviour: cognitive restraint, uncontrolled eating and emotional eating. The items are answered on a 4-point Likert scale. The raw scale scores are transformed to a 0 to 100 scale where higher scores indicate more uncontrolled, restraint and emotional eating.
Change in Systolic and Diastolic Blood pressure | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by measuring the blood pressure.
Change in blood glucose | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by blood test: glucose
Change in blood cholesterol | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by blood test:cholesterol
Change in blood triglycerides | Change from baseline to follow-up at 6-8 months and 12 months.
  Measured by blood test: triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Anderzén Carlsson, RN, Assoc. P, Principal Investigator — Örebro University, Sweden
Locations (1):
- Region Orebro lan, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No